CLINICAL TRIAL: NCT02813720
Title: Distal Phalangeal Bone Involvement Observed by High Resolution Peripheral Quantitative Computed Tomography (HR-pQCT) in Patients With Nail Psoriasis
Brief Title: Distal Erosions and Nail Psoriasis
Acronym: PSUPSO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0202
Record Dates: First submitted 2016-06-22; First posted 2016-06-27 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Psoriatic Arthritis
Keywords: Erosions; Onycholysis; HR-pQCT; Psoriatic arthritis
MeSH Terms: conditions — Arthritis, Psoriatic; Onycholysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine Serum and plasma Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Patients with peripheral PsA
  Interventions: Radiation: HR-pQCT High resolution peripheral quantitative CT-scan
- Patients with psoriatic nail onycholysis
  Interventions: Radiation: HR-pQCT High resolution peripheral quantitative CT-scan
- Patients with PsO only
  Interventions: Radiation: HR-pQCT High resolution peripheral quantitative CT-scan
- Healthy match control subjects
  Interventions: Radiation: HR-pQCT High resolution peripheral quantitative CT-scan

INTERVENTIONS:
Radiation: HR-pQCT High resolution peripheral quantitative CT-scan — HR-pQCT is a powerful device providing low dose irradiation already used in bone field.
  It is a high resolution tool (voxel size=82µm) that the investigators adapted to look after the distal joint involved by onycholysis. An anteroposterior scout view is used to define the region of interest (ROI), which spanned from the top of the distal phalange to the distal part of the intermediate phalange in order to contain the distal joint of the target finger. Images are then analysed for erosions, osteophytes and volumetric bone mineral density.

SUMMARY:
Nearly 30% of patients with cutaneous psoriasis (PsO) developed psoriatic arthritis (PsA). Among these patients 20 % will have severe destructive arthritis. The risk of developing PsA is significantly higher in patients with nail involvement (OR = 2.24; 95% CI [1.26-3.98]). The risk is particularly high for the peripheral form of PsA and onycholysis (OR=2.80; 95% CI [1.34-5.85]).

Thus the investigators wanted to test the hypothesis that onycholysis, in patients without PsA, is a potential clinical marker of subclinical distal enthesopathy and, by extension, of bone micro-structural alterations.

Patients and Methods

The investigators will recruit 4 groups of subjects:

1. Patients with peripheral PsA,
2. Patients with psoriatic nail onycholysis,
3. Patients with PsO only
4. Healthy match control subjects. The investigators will assess the presence of enthesopathy by ultrasonography and bone structural damages (by HR-pQCT) in all subjects at baseline and 4 years.

ELIGIBILITY:
Inclusion Criteria:

* adults over 18 years and until 65 years
* both gender
* covered by the French National Insurance
* subjects entering one of the 4 groups.

Exclusion Criteria:

* Treatment by biological agents are an exclusion criteria for PsO, onycholysis and control patients.
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PSUPSO is a prospective study. Diagnosis of PsA is based on the CASPAR criteria (Taylor 2006). PASI, NAPSI and NAPSI target are recorded. PsO patients are gender and age matched with onycholysis patients patients.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-08 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
distal phalangeal bone erosion of the 2 index fingers of the hand | at baseline and after 4 years of follow-up
  assessment by HR-pQCT

SECONDARY OUTCOMES:
enthesopathy of the 2 index fingers of the hand | at baseline and after 4 years of follow-up
  assessment by ultrasonography
Rheumatoid factors | Biomarkers are assessed at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Cyrille Confavreux, MD PHD, Principal Investigator — Hospices Civils de Lyon, France
Locations (1):
- Centre des Métastases Osseuses (CEMOS) Pavillon F - Rhumatology Hôpital Edouard Herriot, 5 place d'Arsonval, Lyon, France

REFERENCES:
- [Derived] Villani AP, Boutroy S, Coutisson C, Carlier MC, Barets L, Marotte H, Richert B, Chapurlat RD, Jullien D, Confavreux CB. Distal phalangeal bone erosions observed by HR-pQCT in patients with psoriatic onycholysis. Rheumatology (Oxford). 2021 Mar 2;60(3):1176-1184. doi: 10.1093/rheumatology/keaa415. PMID 32885241